CLINICAL TRIAL: NCT00556894
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study of the Safety and Efficacy of Daily CF101 Administered Orally, When Added to Weekly Methotrexate, in Patients With Active Rheumatoid Arthritis
Brief Title: Oral CF101 Tablets and Methotrexate Treatment in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CF101-203RA
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2011-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — CF101; N(6)-(3-iodobenzyl)-5'-N-methylcarboxamidoadenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CF101 0.1 mg (Experimental): CF101 0.1 mg was given orally q12h
  Interventions: Drug: CF101
- CF101 1 mg (Experimental): CF101 1 mg was given orally q12h
  Interventions: Drug: CF101
- Placebo (Placebo Comparator): Matched placebo was given orally q12h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CF101 — orally q12h
  Other Names: IB-MECA
  Arms: CF101 0.1 mg; CF101 1 mg
Drug: Placebo — orally q12h
  Arms: Placebo

SUMMARY:
This trial will test the hypothesis that the addition of CF101, a novel anti-inflammatory agent, will improve the clinical condition of patients with rheumatoid arthritis who still have active joint inflammation despite taking methotrexate for at least 6 months.

DETAILED DESCRIPTION:
This will be a multi-center, randomized, double-blind, parallel-group, placebo-controlled, dose-finding study in which patients with active RA despite receiving methotrexate for at least 6 months (at unchanged doses for >=2 months) will be randomized to the addition of either CF101 0.1 mg, CF101 1 mg, or placebo given orally q12h for 12 weeks. Screening examinations will occur within 1 month prior to dosing. Washout of other disease-modifying antirheumatic drugs (DMARDs) (with the exception of hydroxychloroquine), including biological agents, will occur prior to dosing; if washout is necessary, patients must re-qualify for inclusion following the washout. Doses of nonsteroidal anti-inflammatory drugs (NSAIDS) and corticosteroids must be stable for >=1 month prior to dosing and remain so during protocol participation. Disease activity will be assessed using swollen and tender joint counts, physician and patient global assessments (by visual analog scale, VAS), patient reported pain (by VAS), a Health Assessment Questionnaire (HAQ) Disability Index (DI), Westergren erythrocyte sedimentation rate (ESR, Screening, Weeks 0 and12), and C-reactive protein (CRP) levels. Assessments will take place at Screening, Baseline (Week 0), and at Weeks 2, 4, 8, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18-75 years
* Meet the criteria of the American College of Rheumatology for RA (Arnett FC et al. Arthritis Rheum 1988;31:315-324; refer to Appendix 1. diagnostic criteria for Rheumatoid Arthritis)
* Not bed- or wheelchair-bound
* Active RA, as indicated by the presence of (a) >=6 swollen joints (28 joint count); AND (b) >=6 tender joints (28 joint count); AND either: (c) Westergren ESR of >=28 mm/hour; OR (d) CRP level above the upper limit of normal for the central reference laboratory
* Treatment with weekly oral or parenteral methotrexate for >=6 months prior to baseline
* Methotrexate route of administration has been unchanged for >=2 months prior to baseline
* Dose of methotrexate has been stable at 15-25 mg/week for >=2 months, and is expected to remain stable throughout the study; the stable dose of methotrexate may alternatively be 10-12.5 mg/week if documented toxicity has precluded a higher dose
* If taking hydroxychloroquine or chloroquine, administration duration has been for >=3 months and dose has been stable for >=2 months prior to baseline
* If taking a nonsteroidal anti-inflammatory agent (NSAID), dose has been stable for at least 1 month prior to baseline, and will remain unchanged during protocol participation
* If taking an oral corticosteroid, dose is <10 mg/day prednisone or equivalent, has been stable for at least 1 month prior to the stabilization period, and will remain stable through the stabilization and entire treatment and follow-up period
* Negative screening serum pregnancy test for female patients of childbearing potential
* Females of childbearing potential must utilize, throughout the course of the trial, 2 methods of contraception deemed adequate by the Investigator (for example, oral contraceptive pills plus a barrier method)

Exclusion Criteria:

* Receipt of any of the following for at least a 1 month stabilization period prior to dosing: sulfasalazine, oral or injectable gold, azathioprine, minocycline, penicillamine, anakinra
* Receipt of etanercept for at least a 6 week period prior to dosing
* Receipt of cyclosporine, infliximab or adalimumab for at least a 2 month period prior to dosing
* Receipt of leflunomide for at least a 2 month period prior to screening, unless patient has undergone cholestyramine washout at least 1 month prior to dosing
* Receipt of cyclophosphamide for at least a 6 month period prior to dosing
* Receipt of rituximab at any previous time
* Participation in a previous trial CF101 trial
* Use of oral corticosteroids >10 mg of prednisone, or equivalent, per day
* Change in NSAID dose level for 1 month prior to dosing
* Change in oral corticosteroid dose level during the 1 month prior to, or during, the stabilization period vChange in hydroxychloroquine or chloroquine dose level during the 2 months prior to, or during, the stabilization period
* Receipt of parenteral or intra-articular corticosteroids during the 1 month prior to, or during, the stabilization period
* Significant cardiac arrhythmia or conduction block, congestive heart failure, or any other evidence of clinically significant heart disease; other clinically significant findings on screening electrocardiogram (ECG)
* Hemoglobin level <9.0 gm/dL at the screening visit
* Platelet count <125,000/mm3 at the screening visit
* White blood cell count <3000/mm3 at the screening visit
* Serum creatinine level outside the central laboratory's normal limits at the screening visit
* Liver aminotransferase (ALT and/or AST) levels greater than 1.25 times the central laboratory's upper limit of normal at the screening visit
* Significant acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise patient safety, limit the patient's ability to complete the study, and/or compromise the objectives of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — BioStrategics Consulting Ltd
Locations (26):
- Bulgaria (5):
  - Clinic of Rheumatology at MHAT 'Sveti Georgi', Plovdiv
  - Clinic of Rheumatology at MHAT 'Sveti Ivan Rilski', Sofia
  - Clinic of internal diseases at NMTH 'Tzar Boris Treti', Sofia
  - Second Clinic of Internal Diseases at MHAT 'Stara Zagora', Stara Zagora
  - Clinic of Rheumatology at MHAT 'Sveta Marina' - Varna, Varna
- Czechia (3):
  - University Hospital Hradec Kralove, Hradec Králové
  - Institute of Rheumatology, Prague
  - Rheumotology Out-patient Clinic, Zlín
- Israel (5):
  - Haemek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Rambam Medical Center, Haifa
  - Hadassah Har-Hazofim Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
- Poland (5):
  - Wojewodzki Szpital Zespolony w Elblagu, Elblag
  - Niepubliczny Zaklad Opieki Zdrowotnej, Lublin
  - Wojewodzki Zespol Reumatologiczny w Sopocie, Sopot
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 P.A.M. w Szczecinie, Szczecin
  - Niepubliczny Zaklad Opieki Zdrowotnej "NASZ LEKARZ", Torun
- Serbia (2):
  - Institute of Rheumatology - Belgrade, Belgrade
  - Institute for Prevention, Treatment, and Rehabilitation of Rheumatoid and Cardiovascular Diseases Niska Banja, Niška Banja
- Ukraine (6):
  - Central Municipal Clinical Hospital nº1, Donetsk
  - Kyiv Central Municipal Hospital, Kiev
  - City Clinical Hospital N12, Kiev
  - National Scientific Centre of AMS of Ukraine, Kiev
  - O.O. Bogomolets National Medical University, Kiev
  - Vinnitsya Regional Clinical Hospital, Vinnycia

RESULTS

PARTICIPANT FLOW:
Groups:
- CF101 0.1mg: CF101 0.1mg orally q12 for 12 weeks
- CF101 1mg: CF101 1mg orally q12 for 12 weeks
- Placebo: Matching placebo
Period: Overall Study
Arm/Group | CF101 0.1mg | CF101 1mg | Placebo
Started | 82 | 87 | 84
Completed | 66 | 68 | 65
Not Completed | 16 | 19 | 19
Not completed — Adverse Event | 2 | 3 | 3
Not completed — Death | 1 | 0 | 0
Not completed — regulatory decision in Bulgaria | 10 | 14 | 13
Not completed — Change in therapy | 2 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- CF101 0.1mg; CF101 1mg; Placebo: CF101: orally q12h
- Total: Total of all reporting groups
Arm/Group | CF101 0.1mg | CF101 1mg | Placebo | Total
Number analyzed (Participants) | 82 | 87 | 84 | 253
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 66 | 69 | 69 | 204
  >=65 years | 16 | 18 | 15 | 49
Age, Continuous [Median (Full Range); unit: years] | 55 [24 to 75] | 54 [25 to 75] | 54 [33 to 73] | 54 [24 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 64 | 71 | 203
  Male | 14 | 23 | 13 | 50
Region of Enrollment [Number; unit: participants]
  Serbia | 22 | 20 | 20 | 62
  Ukraine | 22 | 26 | 26 | 74
  Israel | 9 | 9 | 8 | 26
  Bulgaria | 29 | 32 | 30 | 91

OUTCOME MEASURES:

1. Primary Outcome: ACR20 at Week 12
Description: Number of patients that achieved 20% response at week 12 in American College of Rheumatology Criteria
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- CF101 0.1mg: CF101 0.1mg orally q12
- CF101 1mg: CF101 1mg orally q12
- Placebo: Placebo orally q12
Arm/Group | CF101 0.1mg | CF101 1mg | Placebo
Number analyzed (Participants) | 66 | 68 | 65
participants | 29 | 34 | 33

2. Secondary Outcome: ACR 20/50/70, ITT and Evaluable Population, Last Observation Carried Disease Activity Score (DAS28) Change From Baseline at Each Visit in the Efficacy Parameters
Description: ACR20/50/70 responses over time (intent-to-treat [ITT], last observation carried forward [LOCF]), mean changes in individual components of the ACR response criteria, DAS28, European League Against Rheumatism (EULAR) responses
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- CF101 0.1mg: CF101 0.1mg q12 for 12 weeks
- CF101 1mg: CF101 1mg q12 for 12 weeks
- Placebo: Matching Placebo q12 for 12 weeks
Arm/Group | CF101 0.1mg | CF101 1mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/82 | 2/87 | 3/84
Other Adverse Events (participants affected / at risk) | 2/82 | 5/87 | 1/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CF101 0.1mg (N=82) | CF101 1mg (N=87) | Placebo (N=84)
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 — Pancytopenia
Microcytic anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 — HYPOCHROMIC MICROCYTIC ANEMIA III ST.
Alanine aminotransferase and Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 — Elevated ALAT and ASAT
Eyelid oedema (Eye disorders) | 0 | 0 | 1 — OEDEMA OF BOTH EYELIDS WITH CARIAL RASH ON THE NECK
Nausea and Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 — Nausea and Diarrhoea
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CF101 0.1mg (N=82) | CF101 1mg (N=87) | Placebo (N=84)
Nausea (Gastrointestinal disorders) | 2 | 5 | 1 — Nausea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No